CLINICAL TRIAL: NCT01236430
Title: A Study to Evaluate the Definitive Bioequivalence of SCH 900068 With Marketed Products (Protocol No. P07551)
Brief Title: A Study to Determine the Bioequivalence of SCH 900068 Compared to Marketed Products (Protocol No. P07551)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P07551
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; statin; Ezetimibe; Zetia; Atorvastatin; Lipitor
MeSH Terms: conditions — Hyperlipidemias | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ezetimibe 10mg and Atorvastatin 10mg (Active Comparator): Ezetimibe 10mg tablet and Atorvastatin 10mg tablet coadministered
  Interventions: Drug: Ezetimibe; Drug: Atorvastatin 10mg
- 10mg Ezetimibe/10mg Atorvastatin (Experimental): 10mg Ezetimibe/10mg atorvastatin combination tablet
  Interventions: Drug: Ezetimibe/atorvastatin 10mg/10mg FDC
- Ezetimibe 10mg and Atorvastatin 80mg (Active Comparator): Ezetimibe 10mg tablet and Atorvastatin 80mg tablet coadministered
  Interventions: Drug: Ezetimibe; Drug: Atorvastatin 80mg
- 10mg Ezetimibe/80mg Atorvastatin (Experimental): Ezetimibe/atorvastatin 10mg/80mg combination tablet
  Interventions: Drug: Ezetimibe/atorvastatin 10mg/80mg FDC

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 10mg tablet given orally after an overnight fast (at least 10 hours).
  Other Names: Zetia
  Arms: Ezetimibe 10mg and Atorvastatin 10mg; Ezetimibe 10mg and Atorvastatin 80mg
Drug: Ezetimibe/atorvastatin 10mg/10mg FDC — Ezetimibe/atorvastatin 10mg/10mg FDC tablet given orally after an overnight fast (at least 10 hours).
  Other Names: SCH 900068
  Arms: 10mg Ezetimibe/10mg Atorvastatin
Drug: Atorvastatin 10mg — Atorvastatin 10mg given orally after an overnight fast (at least 10 hours).
  Other Names: Lipitor
  Arms: Ezetimibe 10mg and Atorvastatin 10mg
Drug: Atorvastatin 80mg — Atorvastatin 80mg tablet given orally after an overnight fast (at least 10 hours).
  Other Names: Lipitor
  Arms: Ezetimibe 10mg and Atorvastatin 80mg
Drug: Ezetimibe/atorvastatin 10mg/80mg FDC — Ezetimibe/atorvastatin 10mg/80mg FDC tablet given orally after an overnight fast (at least 10 hours).
  Other Names: SCH 900068
  Arms: 10mg Ezetimibe/80mg Atorvastatin

SUMMARY:
The intent of this study is to demonstrate that single doses of the Final Market Image (FMI) ezetimibe/atorvastatin 10mg/10mg and 10mg/80mg fixed dose combination (FDC) tablets are bioequivalent to the same doses of ezetimibe (ZETIA®) and atorvastatin (LIPITOR®) that are coadministered as individual tablets in healthy adults.

ELIGIBILITY:
Inclusion Criteria

* Healthy adult males and females age 18-55 years
* Body mass index (BMI) between 18-35 kg/m^2
* Clinical laboratory tests (complete blood count, blood chemistry, and urinalysis), electrocardiogram, and vital signs must be within normal limits
* Must agree to refrain from consumption of red wine, grapefruit, and grapefruit-containing products, orange and apple juices, and orange- and apple-containing products from beginning approximately 2 weeks prior to administration of the initial dose of study drug, throughout the study (including the washout interval between treatment periods), and until the poststudy visit

Exclusion Criteria

* Female subjects who are pregnant, intend to become pregnant (within 3 months of ending the study), or are nursing/breastfeeding.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug
* History of any infectious disease within 4 weeks prior to drug administration
* Have demonstrated allergic reactions or hypersensitivities or intolerance to atorvastatin or other 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors, ezetimibe, or any component/excipient of the study drug or other food, drug, atopic reactions or asthmatic episodes which, in the opinion of the investigator and sponsor, interfere with their ability to participate in the trial.
* Have a history of prior myopathy or abnormality in liver function studies with statin therapy.
* Are positive for hepatitis B surface antigen, hepatitis C antibodies, or HIV.
* Have donated blood in the past 60 days
* Consume excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time-curve from time zero to infinity (AUC0-∞) of atorvastatin | Hour 0 to Hour 48
Maximum plasma concentration (Cmax) of atorvastatin | Hour 0 to Hour 48
Area under the concentration time-curves from time zero to the time of last measured concentration (AUC0-last) of unconjugated ezetimibe (EZ) | Hour 0 to Hour 96
Maximum plasma concentration (Cmax) of unconjugated ezetimibe (EZ) | Hour 0 to Hour 96

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seiberling, MD, Principal Investigator — Covance Clinical Research Unit AG, Lettenweg 118, CH-4123 Allschwil (Basel), Switzerland